CLINICAL TRIAL: NCT03743428
Title: The Biomarkers Identification for Apatinib and Bevacizumab in the Second-line Therapy for Colorectal Cancer: A Randomised Controlled Trial
Brief Title: Biomarkers for Apatinib and Bevacizumab in Second-line Therapy for Colorectal Cancer(BABST-C)
Acronym: BABST-C
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Too slow speed for recruiting.
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Principal Investigator, Wan He, Professor Wan He, Shenzhen People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Shenzhen CRC-003
Record Dates: First submitted 2018-11-04; First posted 2018-11-16 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Neoplasms
Keywords: apatinib,bevacizumab,FOLFIRI,colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — apatinib; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Head-to-head comparison of apatinib versus bevacizumab plus second-line chemotherapy regimen FOLFIRI for treatment of metastatic colorectal cancer
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib-FOLFIRI (Experimental): Apatinib Mesylate Tablets 250mg po qd Irinotecan 180 mg/m2 IV over 30-90 minutes,day 1 Leucovorin 400 mg/m2 IV infusion to match duration of irinotecan infusion,day 1 5-FU 400 mg/m2 IV bolus day 1,then 1200 mg/m2/d x 2 days (total 2400 mg/m2 over 46-48 hours) continuous infusion Repeat every 2 weeks.
  Interventions: Drug: Apatinib Mesylate Tablets
- Bevacizumab-FOLFIRI (Active Comparator): Bevacizumab Injection 5mg/kg IV,day 1 Irinotecan 180 mg/m2 IV over 30-90 minutes,day 1 Leucovorin 400 mg/m2 IV infusion to match duration of irinotecan infusion,day 1 5-FU 400 mg/m2 IV bolus day 1,then 1200 mg/m2/d x 2days (total 2400 mg/m2 over 46-48 hours) continuous infusion Repeat every 2 weeks.
  Interventions: Drug: Bevacizumab Injection

INTERVENTIONS:
Drug: Apatinib Mesylate Tablets — Apatinib combinated with FOLFIRI regimen as the second-line chemotherapy for mCRC
  Other Names: YN968D1
  Arms: Apatinib-FOLFIRI
Drug: Bevacizumab Injection — Bevacizumab combinated with FOLFIRI regimen as the second-line chemotherapy for mCRC
  Other Names: Avastin
  Arms: Bevacizumab-FOLFIRI

SUMMARY:
Bevacizumab, an antibody against vascular endothelial generated factor (VEGF), combined with the fluorouracil-based chemotherapy regimens has been approved in the 1st and 2nd line treatments for metastatic colorectal cancers(mCRC). Other inhibitors of the VEGF pathway, such as Ramucirumab and Aflibercept are also approved in the 2nd line therapy. Apatinib is a small molecule tyrosine kinase inhibitor (TKI), which can highly selectively bind to and strongly block VEGF receptor 2 (VEGFR - 2), resulting in reduced cell migration, proliferation, and tumor microvascular density mediated by VEGF . In this study, the patients who have progressed following or on the first-line oxaliplatin and fluorouracil（5-FU） combined with bevacizumab are randomised into two arms(FOLFIRI plus apatinib or FOLFIRI plus bevacizumab) in the 2nd line setting. To identify specific biomarkers at the genetic and proteomic levels between two arms is the primary end point.

DETAILED DESCRIPTION:
Based on inclusion and exclusion criteria, eligible mCRC patients are enrolled. the chest-abdonimal-pelvic CT with brain MRI and blood tests are examined to assess base-line measurable lesions and guarantee adequate organ function prior to enrollment. The written consents are signed before enrollment. Randomise patients into two arms: Arm A-apatinib plus FOLFIRI regimen and arm B-bevacizumab plus FOLFIRI regimen. Patients will be given full-dose drugs or reduced-dose drugs if serious toxicities ( CTCAE v4.0 criteria grade 3/4) are complained since previous cycle of treatment.

Symptoms and blood test results (including carcinoembryonic antigen（CEA）and CA199) before each cycle will be recorded. Radiological assessment consisting of chest-abdonimal-pelvic CT together with brain MRI will be performed every 3 months.

Collect biopsy specimens and peripheral blood from mCRC patients every 3 months since randomisation. Identify differential biomarkers between apatinib and bevacizumab and define these biomarkers' prognostic and predictive significances.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable colorectal adenocarcinoma excluding vermiform appendix cancer and anal canal cancer confirmed by histology
* Age ≥18 years ≤ 70 years at the time of informed consent
* Eastern Cooperative Oncology Group（ECOG）performance status (PS) ≤ 1
* Provided informed consent before study-specific screening procedures
* Life expectancy not less than 90 days
* Participants have progressive disease on or within 6 months post the combination of bevacizumab and 5-FU/leucovorin+oxaliplatin(FOLFOX) or capecitabine+oxaliplatin(CAPOX) as the first-line chemotherapy for metastatic colorectal cancer
* Adequate organ function based on the following laboratory values obtained within 14 days prior to enrolment (excluding patients who received blood transfusions or hematopoietic growth factors within 14 days before the laboratory test) Neutrophil count: ≥1500/mm3 Platelet count: ≥10.0 x 104/ mm3 Hemoglobin: ≥9.0 g/dL Total bilirubin: ≤1.5 mg/dL, aspartate aminotransferase (AST), alanine aminotransferase (ALT): ≤100 IU/L (≤200 IU/I if liver metastases present) Serum creatinine: ≤1.5 mg/dL Measurable or nonmeasurable disease based on the Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
* Adequate blood coagulation function [International Normalized Ratio (INR) ≤1.5 and Partial Thromboplastin Time (PTT) or activated PTT (aPTT) ≤1.5 x upper limit of normal (ULN)). Participants on full-dose anticoagulation must be in a stable phase of anticoagulant therapy and if taking oral anticoagulation, participants must have an INR ≤3 without clinically significant active bleeding or a high risk of bleeding
* A historical colorectal cancer tissue sample is available for assessment of biomarkers with signed consent
* Signed informed consent to be provided

Exclusion Criteria:

* History of other malignancy with a disease-free survival <5 years (excluding curatively treated cutaneous basal cell carcinoma, curatively treated cervical in situ carcinoma , and gastroenterological carcinoma confirmed to be cured by endoscopic mucosal resection)
* With a large amount of pleural effusions or ascites requiring intervention
* Radiological evidence of brain metastases or brain tumor
* Actively infectious condition including hepatitis
* One of the following complications: 1) Gastrointestinal obstruction (including paralytic ileus) or gastrointestinal bleeding 2) Symptomatic cardiac disease (including unstable angina, myocardial infarction, and heart failure) 3) Pulmonary fibrosis or interstitial pneumonia 4) Uncontrolled diarrhea (that affects daily activities although adequate therapy 5) Uncontrolled diabetes mellitus
* One of the following medical histories: 1) Myocardial infarction: One episode within one year prior to enrollment or two or more lifetime episodes 2) Remarkable hypersensitivity to any of the study drugs ii) History of side effect to fluoropyrimidines suggestive of dihydropyrimidine dehydrogenase (DPD) deficiency
* Pregnant or lactating females, and males and females reluctant to use contraception
* Psychiatric disability that would disturb study compliance
* Other conditions determined by the investigator to be not suitable for participation in the study
* History of concurrent gastrointestinal perforation or gastrointestinal perforation within 1 year prior to enrollment
* Pulmonary hemorrhage/hemoptysis ≥ Grade 2 (identified as bright red blood of not less 2.5mL) within 1 month before enrollment.
* History of thoracotomy,laparotomy, or intestinal resection within 28 day prior to enrollment
* Unhealed wound (other than suture wounds due to implantation of a central venous port), traumatic fracture, or gastrointestinal ulcer
* Current cerebrovascular disease or thromboembolism or either within 1 year before enrollment
* Current anticoagulation therapy or requiring anticoagulation agents (> 325 mg/day of aspirin)
* Bleeding diathesis, coagulopathy, or coagulation factor abnormality (INR

  ≥1.5 within 14 days before enrollment)- Page 6 of 7 [DRAFT] -
* Uncontrolled hypertension Urine dipstick for proteinuria >+2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify biomarkers specific to apatinib or bevacizumab by transcriptome analysis | 4 years
  Identify differentially expressed genes specific to apatinib or bevacizumab by the next-generation RNA-seq technology .
Identify biomarkers specific to apatinib or bevacizumab by proteomic analysis | 4 years
  Identify proteomic molecules specific to apatinib or bevacizumab by the photoreactive crosslinking, pull-down, affinity purification and mass spectrometry (AP-MS) analyses

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | The follow-up period ranges from the first patient recruited to the last patient within 6 months after admission, up to 2 years
  PFS was defined as the time from the date of randomization until the date of objectively determined progressive disease (PD) [according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v). 1.1] or death due to any cause, whichever was first. PD is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). Participants who died without a reported prior progression were considered to have progressed on the day of their death. Participants who did not progress or were lost to follow-up were censored at the day of their last radiographic tumor assessment.
Overall Survival (OS) | The follow-up period ranges from the first patient recruited to the last patient within 6 months after admission,up to 2 years
  OS was defined as the time in months from the date of randomization to the date of death from any cause. For participants not known to have died as of the cut-off date, OS was censored at the last known date alive.

CONTACTS AND LOCATIONS:
Overall Officials: Wan He, PhD,MD, Principal Investigator — Shenzhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

REFERENCES:
- [Background] Bennouna J, Sastre J, Arnold D, Osterlund P, Greil R, Van Cutsem E, von Moos R, Vieitez JM, Bouche O, Borg C, Steffens CC, Alonso-Orduna V, Schlichting C, Reyes-Rivera I, Bendahmane B, Andre T, Kubicka S; ML18147 Study Investigators. Continuation of bevacizumab after first progression in metastatic colorectal cancer (ML18147): a randomised phase 3 trial. Lancet Oncol. 2013 Jan;14(1):29-37. doi: 10.1016/S1470-2045(12)70477-1. Epub 2012 Nov 16. PMID 23168366
- [Background] Van Cutsem E, Tabernero J, Lakomy R, Prenen H, Prausova J, Macarulla T, Ruff P, van Hazel GA, Moiseyenko V, Ferry D, McKendrick J, Polikoff J, Tellier A, Castan R, Allegra C. Addition of aflibercept to fluorouracil, leucovorin, and irinotecan improves survival in a phase III randomized trial in patients with metastatic colorectal cancer previously treated with an oxaliplatin-based regimen. J Clin Oncol. 2012 Oct 1;30(28):3499-506. doi: 10.1200/JCO.2012.42.8201. Epub 2012 Sep 4. PMID 22949147
- [Background] Tabernero J, Yoshino T, Cohn AL, Obermannova R, Bodoky G, Garcia-Carbonero R, Ciuleanu TE, Portnoy DC, Van Cutsem E, Grothey A, Prausova J, Garcia-Alfonso P, Yamazaki K, Clingan PR, Lonardi S, Kim TW, Simms L, Chang SC, Nasroulah F; RAISE Study Investigators. Ramucirumab versus placebo in combination with second-line FOLFIRI in patients with metastatic colorectal carcinoma that progressed during or after first-line therapy with bevacizumab, oxaliplatin, and a fluoropyrimidine (RAISE): a randomised, double-blind, multicentre, phase 3 study. Lancet Oncol. 2015 May;16(5):499-508. doi: 10.1016/S1470-2045(15)70127-0. Epub 2015 Apr 12. PMID 25877855
- [Background] Fuchs CS, Tomasek J, Yong CJ, Dumitru F, Passalacqua R, Goswami C, Safran H, Dos Santos LV, Aprile G, Ferry DR, Melichar B, Tehfe M, Topuzov E, Zalcberg JR, Chau I, Campbell W, Sivanandan C, Pikiel J, Koshiji M, Hsu Y, Liepa AM, Gao L, Schwartz JD, Tabernero J; REGARD Trial Investigators. Ramucirumab monotherapy for previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (REGARD): an international, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2014 Jan 4;383(9911):31-39. doi: 10.1016/S0140-6736(13)61719-5. Epub 2013 Oct 3. PMID 24094768
- [Background] Wilke H, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Sugimoto N, Lipatov O, Kim TY, Cunningham D, Rougier P, Komatsu Y, Ajani J, Emig M, Carlesi R, Ferry D, Chandrawansa K, Schwartz JD, Ohtsu A; RAINBOW Study Group. Ramucirumab plus paclitaxel versus placebo plus paclitaxel in patients with previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (RAINBOW): a double-blind, randomised phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1224-35. doi: 10.1016/S1470-2045(14)70420-6. Epub 2014 Sep 17. PMID 25240821
- [Background] Garon EB, Ciuleanu TE, Arrieta O, Prabhash K, Syrigos KN, Goksel T, Park K, Gorbunova V, Kowalyszyn RD, Pikiel J, Czyzewicz G, Orlov SV, Lewanski CR, Thomas M, Bidoli P, Dakhil S, Gans S, Kim JH, Grigorescu A, Karaseva N, Reck M, Cappuzzo F, Alexandris E, Sashegyi A, Yurasov S, Perol M. Ramucirumab plus docetaxel versus placebo plus docetaxel for second-line treatment of stage IV non-small-cell lung cancer after disease progression on platinum-based therapy (REVEL): a multicentre, double-blind, randomised phase 3 trial. Lancet. 2014 Aug 23;384(9944):665-73. doi: 10.1016/S0140-6736(14)60845-X. Epub 2014 Jun 2. PMID 24933332